CLINICAL TRIAL: NCT03022201
Title: Therapeutic Efficacy of DA-9701 on Gastric Motility in Patients With Parkinson's Disease Evaluated by Magnetic Resonance Imaging: A Randomized Controlled, Double-Blind, Non-Inferiority Trial
Brief Title: Comparing the Therapeutic Efficacy and Safety of DA-9701 With Domperidone in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1210/173-006
Record Dates: First submitted 2016-11-23; First posted 2017-01-16 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2017-01

CONDITIONS: Parkinson's Disease,Idiopathic
Keywords: Motilitone
MeSH Terms: conditions — Parkinson Disease | interventions — DA-9701; Domperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-9701 (Experimental): In this arm, the study participants will receive DA-9701 30mg + placebo domperidone tablet tid ac for 4 weeks.
  Interventions: Drug: DA-9701; Drug: Placebo domperidone
- Domperidone (Active Comparator): (This study is a randomized, double-blinded, non-inferiority trial. Thus it is designed to have no placebo arm.) In this arm, the study participants will receive domperidone 10mg + placebo DA-9701 tablet tid ac +for 4 weeks.
  Interventions: Drug: Domperidone; Drug: Placebo DA-9701

INTERVENTIONS:
Drug: DA-9701 — Following 2-week screening period, study participants in this group will be given a standard dose of DA-9701 (30 mg t.i.d). Concomitant anti-PD medication will be continued without modification during the trial. The investigators will evaluate dyspepsia and constipation symptoms, gastric emptying by MRI, UPDRS and clinical variables at baseline and at the end of the study.
  Other Names: Motilitone
  Arms: DA-9701
Drug: Domperidone — Following 2-week screening period, study participants in this group will be given a standard dose of domperidone (10 mg t.i.d). Concomitant anti-PD medication will be continued without modification during the trial. The investigators will evaluate dyspepsia and constipation symptoms, gastric emptying by MRI, UPDRS and clinical variables at baseline and at the end of the study.
  Other Names: Motilium-M
  Arms: Domperidone
Drug: Placebo domperidone
  Arms: DA-9701
Drug: Placebo DA-9701
  Arms: Domperidone

SUMMARY:
This study will evaluate the therapeutic efficacy and safety of DA-9701 with domperidone in patients with Parkinson's disease

DETAILED DESCRIPTION:
To prevent nausea and vomiting induced by anti-parkinsonian drugs, prokinetic drugs are frequently prescribed in patients with Parkinson's disease (PD). Additionally, there has been some evidence that prokinetics might improve PD symptom fluctuations. From this background, the investigators will evaluate the therapeutic efficacy and safety of DA-9701 in PD patients.

In this study, 40 patients will be enrolled and randomly allocated 1:1 to receive either domperidone or DA-9701. The gastric function of each study participant will be evaluated using the MRI technique before and after 4 weeks of the treatment. The study participants will also be subjected to complete the gastrointestinal symptom diary before and during the treatment period. In addition, plasma levodopa concentrations will be determined 30 minutes after dose administration before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* subjects diagnosed with spontaneous parkinsonism by the United Kingdom(UK) Parkinson's Disease Society Brain Bank criteria
* subjects who are able to explain symptoms they experience and to complete relevant assessment and exams including questionaires
* subjects who understand the purpose and protocols of the study and agree to participate on the study

Exclusion Criteria:

* subjects who experience psychiatrical disorders such as cognitive or behavioral disorders
* subjects who are on prokinetics or who are unable to cease such medication
* subjects who present neurological disorders which influence gastrointestinal mobility
* subjects who present gastrointestinal conditions which influence gastrointestinal mobility
* subjects with a history of gastrectomy or colectomy
* subjects who are unable to receive and complete the course of medication due to other metabolic disorders
* subjects diagnosed with parkinson plus syndrome
* subjects who are unable to undergo MRI scan for safety reasons due to claustrophobia or certain devices such as cardiac pacemakers or aneurysm clips

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change of gastric motility evaluated using MRI from baseline at 4 weeks after the treatment | 0, 4 weeks
  MRI is known to be accurate and useful in evaluating gastric motility. Gastric emptying rate (GER) evaluated using MRI will be compared before and after the treatment, and between the groups.

SECONDARY OUTCOMES:
Patient's symptoms of dyspepsia and constipation assessed patient diary | -1 to 4 weeks
  The study participants will fill up the gastrointestinal symptom diary before and during the treatment period. In addition, the investigators will assess the Patient's Global Assessment (PGA) for dyspeptic symptoms at the end of the treatment period.
Levodopa plasma concentration 30 minutes after the L-dopa administration | 0, 4 weeks
  Plasma levodopa concentrations will be determined 30 minutes after L-dopa dose administration before and after treatment.
UPDRS Part III score | 0, 4 weeks
  To evaluate any deteriorations in Parkinson's disease, the investigators will assess Unified Parkinson's Disease Rating Scale (UPDRS) score before and after treatment in the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Min Shin, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Cheol Min Shin, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin CM, Lee YJ, Kim JM, Lee JY, Kim KJ, Choi YJ, Kim N, Lee DH. DA-9701 on gastric motility in patients with Parkinson's disease: A randomized controlled trial. Parkinsonism Relat Disord. 2018 Sep;54:84-89. doi: 10.1016/j.parkreldis.2018.04.018. Epub 2018 Apr 21. PMID 29705555